CLINICAL TRIAL: NCT01258465
Title: Research in Autism: Parent Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Laura Schreibman, Ph.D., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH39434
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Autistic Disorder
Keywords: Communication; Pivotal Response Training; Picture Exchange Communication System
MeSH Terms: conditions — Autistic Disorder; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pivotal Response Training (Active Comparator): A naturalistic behavioral intervention designed to facilitate verbal communication.
  Interventions: Behavioral: Pivotal Response Training; Behavioral: Picture Exchange Communication System
- Picture Exchange Communication System (Active Comparator): Pictorially-based behavioral protocol designed to facilitate communication via picture icons.
  Interventions: Behavioral: Picture Exchange Communication System

INTERVENTIONS:
Behavioral: Pivotal Response Training — Naturalistic behavioral protocol designed to teach vocal communication.
  Arms: Pivotal Response Training
Behavioral: Picture Exchange Communication System — Pictorially-based behavioral protocol designed to teach communication to nonverbal children via pictures icons.

SUMMARY:
The purpose of this research project was to systematically compare two widely used types of intervention programs for children with autism within a parent training model. In one condition, randomly assigned children were provided with an intervention that typically results in acquisition of expressive words in a large percentage of children diagnosed as having autism, using a well-documented manualized intervention focused on verbal expressive communication only (Pivotal Response Training, PRT). In the other condi¬tion, randomly assigned children received a widely used intervention on the same social communication functions using a well-documented manualized augmentative system of intervention (Picture Exchange Communica¬tion System, PECS) that has been reported to produce verbal and nonverbal communication in large percentages of children diagnosed with autism. Children in the two conditions were compared for development of verbal and nonverbal communication, changes in disruptive behavior, changes in symptoms of autism, and general adaptive behavior gains. In addition, parent satisfaction and stress measures were gathered in order to assess the effects of each intervention on family functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autistic Disorder or At Risk of Autistic Disorder
* Age 2-0 to 3-11 years of age
* Use of fewer than 10 functional words at intake

Exclusion Criteria:

* Primary diagnosis of mental retardation
* Neurologic pathology (e.g., PKU, encephalitis, brain trauma)
* Major sensory impairment

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mullen Scales of Early Learning | 23 weeks with three months follow-up

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales | 23 weeks and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Schreibman, Ph.D., Principal Investigator — University of California, San Diego; Robert L Koegel, Ph.D., Principal Investigator — University of California, Santa Barbara
Locations (2):
- United States (2):
  - University of California, San Diego Psychology Department, La Jolla, California
  - University of California, Santa Barbara, School of Education, Department of Clinical, Counseling, and School Psychology, Santa Barbara, California